CLINICAL TRIAL: NCT06024642
Title: Multicenter, Randomized, Double-blind Placebo-controlled, Crossover Study to Investigate Effects of V117957 in Female Subjects With Overactive Bladder Syndrome
Brief Title: Study of V117957 in Overactive Bladder Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imbrium Therapeutics (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OAG1030
Record Dates: First submitted 2023-08-17; First posted 2023-09-06 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V117957 (Experimental)
  Interventions: Drug: V117957
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V117957 — V117957 1 mg - 1 tablet taken orally at bedtime.
  Other Names: Sunobinop
  Arms: V117957
Drug: Placebo — Placebo to match V117957 tablets - 1 tablet taken orally at bedtime.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of V117957 in subjects with overactive bladder syndrome, compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria include:

1. Female, age ≥18-70 years and capable of voiding independently. Able to comply with acceptable methods of contraception.
2. Has symptoms of overactive bladder including (OAB) urinary urgency and urinary frequency with incontinence for ≥3 months.
3. Willing to modify current OAB treatment regimen.

Key Exclusion Criteria include:

1. Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor.
2. Urinary tract infection (UTI) within past 30 days, or history of recurrent UTI.
3. Hematuria associated with bladder malignancy or other significant pathology.
4. Had surgical procedure that affected bladder function.
5. Received intravesical therapy within past 12 months or had bladder hydrodistention within past 6 months.
6. Grade III/IV pelvic organ prolapse with/without cystocele or urethral diverticulum.
7. Clinically significant kidney disease or nephrolithiasis.

Other protocol-specific inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Arizona Urology Specialists, PLLC, Tucson, Arizona
  - Hope Clinical Research, LLC, Canoga Park, California
  - ARK Clinical Research, Long Beach, California
  - Urology Group of Southern California, Los Angeles, California
  - Providea Health Partners, LLC, Evergreen Park, Illinois
  - DelRicht Research, New Orleans, Louisiana
  - Ochsner LSU Health Shreveport - Regional Urology, Shreveport, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - AccuMed Research Associates, Garden City, New York
  - Unified Women's Clinical Research-Lyndhurst, Winston-Salem, North Carolina
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center translational study conducted at study sites in the US.
Pre-assignment Details: This was a two-period single-sequence crossover design with investigative sites and subjects blinded to both the randomization eligibility criteria and the assignment of subjects to only a single treatment sequence (placebo followed by active). The study included a single-blind run-in phase (2-week placebo exposure); a double-blind treatment phase (2-weeks placebo immediately followed by 6-weeks V117957 exposure); and a safety follow-up phase (2 weeks duration).
Groups:
- All Study Participants: Placebo for 2 weeks (single-blind run-in), then placebo for 2 weeks immediately followed by V117957 for 6 weeks (double-blind treatment phase) then placebo for 1 week (safety follow-up phase).
Period: Single-blind Run-in Period
Arm/Group | All Study Participants
Started | 51
Completed | 51
Not Completed | 0
Period: Double-blind / Safety Follow-up Phase
Arm/Group | All Study Participants
Started | 51 (One subject was randomized but did not receive study drug.)
Completed | 47
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: The group of subjects who were randomized and received at least 1 dose of study drug during the double-blind treatment phase.
Arm/Group | All Study Participants
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 33
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Micturition Episode Components (Micturition, Incontinence, and Urgency) Per 24 Hours.
Description: Subjects were asked to record all micturition episode components into a daily electronic diary during the 3 to 7 days prior to each scheduled clinic visit.
Time Frame: Baseline, Weeks 2, and 8
Population: The full analysis population is the group of subjects who were randomized, received study drug, and had at least 1 valid efficacy measurement.
Measure: Mean (Standard Deviation); unit: Episodes per 24 hours
Groups:
- Week 2 (Placebo): Placebo for 2 weeks.
- Week 8 (V117957): V117957 for 6 weeks.
Arm/Group | Week 2 (Placebo) | Week 8 (V117957)
Number analyzed (Participants) | 47 | 44
Episodes per 24 hours
  Number of Micturition Episodes per 24 hours | -0.8 (1.97) | -0.8 (2.32)
  Number of Incontinence Episodes per 24 hours: number analyzed (Participants) | 43 | 41
  Number of Incontinence Episodes per 24 hours | -0.2 (0.60) | -0.4 (0.81)
  Number of Urgency Episodes per 24 hours | -0.5 (1.20) | -0.5 (2.07)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported starting from the time informed consent for study participation was provided up to 16 weeks. All-cause mortality and serious adverse events were reported from the start of study participation up to 30 days after last study drug dose (approximately 20 weeks).
Groups:
- Single-blind Run-in Period (Placebo); Double-blind Treatment Phase (Placebo): Placebo for 2 weeks.
- Double-blind Treatment Phase (V117957): V117957 for 6 weeks.
- Safety Follow-up Phase (Placebo): Placebo for 1 week.
Arm/Group | Single-blind Run-in Period (Placebo) | Double-blind Treatment Phase (Placebo) | Double-blind Treatment Phase (V117957) | Safety Follow-up Phase (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50 | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/48 | 1/47
Other Adverse Events (participants affected / at risk) | 3/51 | 1/50 | 6/48 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-blind Run-in Period (Placebo) (N=51) | Double-blind Treatment Phase (Placebo) (N=50) | Double-blind Treatment Phase (V117957) (N=48) | Safety Follow-up Phase (Placebo) (N=47)
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-blind Run-in Period (Placebo) (N=51) | Double-blind Treatment Phase (Placebo) (N=50) | Double-blind Treatment Phase (V117957) (N=48) | Safety Follow-up Phase (Placebo) (N=47)
Urinary tract infection (Infections and infestations) | 3 | 1 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT06024642/Prot_SAP_000.pdf